CLINICAL TRIAL: NCT00086333
Title: A Phase II Study Using FDG-PET to Investigate the Dosing Schedule and Response of Combination SGN-15 (cBR96-Doxorubicin Immunoconjugate) and Docetaxel in Patients With Stage IV or Stage IIIB Non-Small Cell Lung Carcinoma Ineligible for Combined Modality Treatment With Curative Intent
Brief Title: FDG-PET to Investigate SGN-15 and Docetaxel in Patients With Advanced Non-Small Cell Lung Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SG015-0005
Record Dates: First submitted 2004-06-30; First posted 2004-07-02 (Estimated); Last update posted 2011-10-24 (Estimated); Status verified 2011-10

CONDITIONS: Non-Small Cell Lung Carcinoma
Keywords: Carcinoma, Non-Small-Cell Lung; Taxotere; docetaxel; taxanes
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel

INTERVENTIONS:
Drug: SGN-15, Docetaxel

SUMMARY:
This is an open-label, randomized phase II trial of a monoclonal antibody (mAb) drug immunoconjugate, SGN-15, administered weekly in combination with weekly docetaxel. The primary objective of the study is to determine the optimal interval between SGN-15 and docetaxel using FDG-PET imaging as a surrogate marker of response. In addition, clinical response rate, duration of response, and survival data will be collected.

DETAILED DESCRIPTION:
SGN-15 is a mAb-drug immunoconjugate comprised of the chimeric anti-Lewis Y (LeY) mAb BR96, conjugated to doxorubicin. The LeY antigen is found as a glycoprotein at the cell surface on 90% of carcinomas of the lung. SGN-15 induces its antitumor effect through binding to the cell surface LeY antigen. It is then rapidly internalized with release of doxorubicin inside the cell allowing the relative sparing of tissues normally affected by non-specific chemotherapy.

The study is open to patients with good performance status (ECOG 0<=2) with stage IIIB or IV NSCLC which is not potentially curable by surgery or combined modality therapy and who have received no prior lung cancer chemotherapy for metastatic NSCLC.

Patients will be registered into one of two treatment sequences and wil receive SGN-15 and docetaxel in 4 week cycles consisting of treatment weekly for 3 weeks, followed by a week of rest.

Arm A will receive a combination os SGN-15 and docetaxel on the same day. Arm B will receive the combination of SGN-15 followed by the docetaxel 3 days later. All patients will undergo PET imaging prior to treatment and on Day 22.

Patients achieving a clinical response or stable disease as determined by physical examination and/or traditional restaging studies (using established RECIST criteria) after one 4 week cycle of therapy are eligible to receive continued cycles of SGN-15 and docetaxel on the same schedule until clinical or radiographic disease progression or toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically confirmed stage IIIB or IV NSCLC with a minimum of 1 measurable baseline target lesion who have received no prior chemotherapy for metastatic disease and are not eligible for combined modality therapy with curative intent
* Patients must have an ECOG performance status of less than or equal to 2
* -Patients must have a tumor block available for documentation of LeY antigen expression by immunohistochemistry
* -FDG-PET imaging must be completed at a PET center approved by Seattle Genetics
* Patients must have adequate bone marrow and hepatic function

Exclusion Criteria:

* -Prior cytotoxic therapy for metastatic NSCLC
* -Those with serious underlying non-malignant disease
* -Patients with peripheral neuropathy > Grade 2 are excluded from study
* -Patients with IDDM or NIDDM
* Patients with known active viral, bacterial, or symptomatic fungal infection
* Concomitant with other antineoplastic or experimental agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-07; Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Chicago, Chicago, Illinois
  - The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Providence Health System, Regional Cancer Program, Portland, Oregon
  - Kaiser Permanente, Portland, Oregon